CLINICAL TRIAL: NCT05263557
Title: Dissecting the IMpact of 11-OXygenated and Classic Androgens on Skeletal Muscle Insulin Sensitivity (DIMOXIS)
Acronym: DIMOXIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University of Oxford (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DIMOXIS
Record Dates: First submitted 2021-10-20; First posted 2022-03-02 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance; Androgen; Hypersecretion; Endocrine System Diseases
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Endocrine System Diseases | interventions — Dehydroepiandrosterone; adrenosterone

STUDY DESIGN:
Intervention Model Description: Interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHEA (Experimental): Adult females with polycystic ovary syndrome (PCOS) and evidence of clinical or biochemical androgen excess will be recruited and randomised.
  Interventions: Dietary Supplement: Dehydroepiandrosterone (DHEA)
- 11KA4 (Experimental): Adult females with polycystic ovary syndrome (PCOS) and evidence of clinical or biochemical androgen excess will be recruited and randomised.
  Interventions: Dietary Supplement: 11-ketoandrostenedione (11KA4)

INTERVENTIONS:
Dietary Supplement: Dehydroepiandrosterone (DHEA) — Dehydroepiandrosterone (DHEA) at a dose of 150mg once daily for 7 days.
  Arms: DHEA
Dietary Supplement: 11-ketoandrostenedione (11KA4) — 11ketoandrostenedione (11KA4) at a doses of 150mg once daily for 7 days.
  Arms: 11KA4

SUMMARY:
Androgen excess is the cardinal biochemical feature of polycystic ovary syndrome (PCOS). Serum testosterone correlates with insulin resistance in PCOS, however, there is an urgent need to improve our understanding of the association between androgens and the risk of type 2 diabetes.

11-oxygenated steroids are the predominant androgens in PCOS and correlate closely with markers of insulin resistance. The bioactive 11-oxygenated androgen 11-ketotestosterone (11KT) binds and activates the androgen receptor with equal affinity to testosterone, yet nothing is known about its impact on metabolism or glucose homeostasis

Crucially, there are no data linking androgen excess with muscle glucose metabolism and the differential contribution of 11-oxygenated androgens to diabetes risk through these processes remains unknown.

The investigators hypothesise the following:

1. Oral androgen exposure in women with PCOS results in distinct changes in tissue-specific insulin sensitivity and muscle energy biogenesis
2. 11-oxygenated androgen exposure exerts differential changes on the above parameters in comparison to classic androgen exposure

The study has the following aims:

1. To examine the impact of oral androgen exposure on skeletal muscle insulin sensitivity and glucose disposal in women with PCOS.
2. To delineate the impact of androgen exposure on muscle mitochondrial function ex vivo in women with PCOS
3. To compare the differential impact of 11-oxygenated androgen compared to classic androgens on glucose disposal and muscle mitochondrial function

The two arms will run in parallel and all participants will undergo identical investigations before and after 7 days of either DHEA or 11KA4.

Investigations will include baseline arthrometric measurements muscle biopsy, two-step hyperinsulinaemic euglycaemic clamp, breath sampling.

This interventional metabolic phenotyping study will probe the role of classic and 11-oxygenated androgens in metabolic dysfunction in PCOS using gold-standard in vivo metabolic phenotyping techniques. Delineating the distinct contribution of 11-oxygenated androgens, through effects on skeletal muscle biology, to the risk of T2DM is an important step in the process of determining risk of type 2 diabetes in this vulnerable cohort.

ELIGIBILITY:
Inclusion Criteria:

* Women with a confirmed diagnosis polycystic ovary syndrome with androgen excess on clinical or biochemical grounds
* BMI 20.0-39.9kg/m2
* Age range 18-40 years
* Ability to provide informed consent

Exclusion Criteria:

* A confirmed diagnosis of diabetes
* Current or recent (<3-months) use of weight loss medications
* Current or recent use of oral contraceptive pill or hormone replacement therapy (within 3-months)
* Blood haemoglobin <12.0g/dL
* History of alcoholism or a greater than recommended alcohol intake (recommendations > 21 units on average per week for men and > 14 units on average per week for women)
* Haemorrhagic disorders or Treatment with anticoagulant agents
* Any medical condition in the opinion of the investigator that might impact upon safety or validity of the results
* Pregnancy or breastfeeding at the time of planned recruitment
* A diagnosis of PCOS according to Rotterdam criteria where the patient does not have clinical or biochemical evidence of androgen excess
* History of significant renal (eGFR<30) or hepatic impairment (AST or ALT >two-fold above ULN; pre-existing bilirubinaemia >1.2 ULN)
* Any other significant disease or disorder that, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Current intake of drugs known to impact upon steroid or metabolic function or intake of such drugs during the six months preceding the planned recruitment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Relative change in glucose disposal from baseline with 11KA4 administration compared to that seen with DHEA | 7 Days
  Utilizing hyperglycaemic-euglycaemic clamp (μmol/min/kg)

SECONDARY OUTCOMES:
Relative change in glucose oxidation from baseline with 11KA4 administration compared to that seen with DHEA | 7 Days
  Measured by 13C-breath testing (mg/kg/min)
Relative change in endogenous glucose production from baseline with 11KA4 administration compared to that seen with DHEA (μmol/min/kg) | 7 Days
  Utilizing hyperglycaemic-euglycaemic clamp (μmol/min/kg)

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Michael, Principal Investigator — RCSI Education & Research Centre, Beaumont Hospital, Beaumont Dublin 9 Ireland Ireland
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No